CLINICAL TRIAL: NCT00540020
Title: Rehabilitation of Traumatic Brain Injury in Active Duty Military Personnel and Veterans: DVBIC Randomized Clinical Trial of Two Rehabilitation Approaches
Brief Title: Rehabilitation of Traumatic Brain Injury in Active Duty Military Personnel and Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Collaborators: James A. Haley Veterans Administration Hospital (U.S. Federal Agency); Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F292BL-C9; F292BL-C8; F292BL-C7; F292BL-C6
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injuries; Cognition; Randomized Trials; Rehabilitation; Treatment Outcome
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Cognitive-Didactic (Experimental): Developed by Sohlberg & Mateer to target four cognitive domains often impaired by TBI: attention, memory, executive functions, and pragmatic communication. Subjects practiced progressively more difficult paper-and-pencil or computerized cognitive tasks in 1:1 cognitive therapy sessions (1.5-2.5 hours daily).
  Interventions: Other: Rehabilitation
- Functional-Experiential (Experimental): The works of Giles and Clark-Wilson and Hartley guided the basic concepts and treatment of the functional-experiential arm (Functional). The objective of the functional protocol was to use real life performance situations and common tasks to remediate or compensate for functional deficits after brain injury. Functional protocol treatment interventions (1.5-2.5 hours daily) typically occurred in group settings and natural environments (hospital recreation areas, group rooms, simulated home environments in the dining room, community outings, etc.).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation

SUMMARY:
Context: Traumatic brain injury (TBI) is a common condition associated with significant long-term cognitive, behavioral, and functional morbidities. There are minimal controlled efficacy data of various acute rehabilitation intervention approaches.

Objective: To determine the relative efficacy of two different acute TBI rehabilitation approaches - cognitive-didactic versus functional-experiential. Secondarily to determine relative efficacy for different patient subpopulations based on baseline cognitive functioning.

DETAILED DESCRIPTION:
A randomly assigned, intent-to-treat model of two different comprehensive treatment programs conducted between July 19 1996 and May 16, 2003 in 360 adult participants with moderate to severe TBI treated in four participating Veterans Administration TBI rehabilitation centers.

All patients admitted to the Commission for Accreditation of Rehabilitation Facilities (CARF) accredited acute inpatient rehabilitation brain injury programs at 4 participating Veterans Administration Medical Centers (VAMCs) (Minneapolis, Palo Alto, Richmond, and Tampa) during the study enrollment period were screened for eligibility.

The design was a randomized-controlled trial with two treatment arms (cognitive-didactic and functional-experiential), both embedded within an interdisciplinary TBI rehabilitation program. All treatment was hospital based. The interactive nature of the experimental conditions precluded subject blinding. Since each participating site serves a wide geographic area, the protocol permitted post-hospital outcome assessments by structured telephonic interview, to minimize drop out.

Participants completed baseline assessment then received by random assignment one of the two standardized protocol rehabilitation programs (summarized below and described in detail elsewhere). Participants received 1.5 to 2.5 hours daily of protocol-specific therapy plus another 2 to 2.5 hours daily of occupational and physical therapy. Independent teams of therapists functioned at each site to deliver the separate treatments and by necessity were not blinded to treatment. Protocol monitoring site visits, biweekly conference calls, and biannual investigator meetings were conducted to ensure uniformity of protocol treatment over time.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe closed head injury, manifested by a post-resuscitation Glasgow Coma Scale (GCS) score of 12 or less, or coma of 12 hours or more , or posttraumatic amnesia (PTA) of 24 hours or more, and/or focal cerebral contusion or hemorrhage on computed tomography (CT) or magnetic resonance imaging (MRI)
* documented traumatic brain injury within 6 months of randomization
* Rancho Los Amigos Scale (RLAS) cognitive level of 5-7 at time of randomization
* age 18 or older
* active duty military member or veteran
* anticipated length of needed acute interdisciplinary TBI rehabilitation of 30 days or more

Exclusion Criteria:

* history of prior moderate to severe traumatic brain injury or other pre-injury severe neurologic or psychiatric condition, such as psychosis, stroke, multiple sclerosis, or spinal cord injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 1996-07; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
(1) Functional independence (i.e., ability to live independently with less than 3 hours of assistance per week) (2) Return to work/school (i.e., paid employment or school enrollment, either full or part time) | One-year Follow-up

SECONDARY OUTCOMES:
The Functional Independence Measures (FIM)33, 34 consisting of motor and cognitive scores and the Disability Rating Scale Score (DRS)35 were measured. | Discharge from Protocol Treatment
Quality of life, psychosocial function, behavioral, and mood state measures | One-year Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Warden, M.D., Principal Investigator — The Defense and Veterans Brain Injury Center; Elaine Date, M.D., Principal Investigator — VA Palo Alto Health Care System; Steven Scott, D.O., Principal Investigator — James A. Haley VA; Barbara Sigford, M.D., Ph.D., Principal Investigator — Minneapolis VA; William Walker, M.D., Principal Investigator — Hunter H. McGuire VAMC

REFERENCES:
- [Derived] Vanderploeg RD, Schwab K, Walker WC, Fraser JA, Sigford BJ, Date ES, Scott SG, Curtiss G, Salazar AM, Warden DL; Defense and Veterans Brain Injury Center Study Group. Rehabilitation of traumatic brain injury in active duty military personnel and veterans: Defense and Veterans Brain Injury Center randomized controlled trial of two rehabilitation approaches. Arch Phys Med Rehabil. 2008 Dec;89(12):2227-38. doi: 10.1016/j.apmr.2008.06.015. PMID 19061734